CLINICAL TRIAL: NCT03379415
Title: The Effect of Commercially Available Footwear Interventions on Biomechanical Outcomes Associated With Knee Osteoarthritis in Meniscectomy Patients
Brief Title: The Effect of Commercially Available Footwear Interventions in Meniscectomy Patients
Acronym: MENI-FOOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salford (Other)
Responsible Party: Principal Investigator, Vanessa Walters, Principal Investigator, University of Salford
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSR1617-140
Record Dates: First submitted 2017-11-20; First posted 2017-12-20 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Meniscus Injury; Osteoarthritis, Knee; Footwear
Keywords: Meniscectomy; Footwear; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Gait Analysis

STUDY DESIGN:
Intervention Model Description: Testing meniscus patients for several different shoes
Who Masked: Participant
Masking Description: Only the participant is blinded to the randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meniscus Injured (Experimental): These meniscus patients will be recruited to participate in a single session to wear 4 different pairs of shoes
  Interventions: Device: Footwear
- Footwear (Experimental): 4 Different types of trainers will be used to see the difference in gait in meniscectomy patients
  Interventions: Procedure: Gait analysis

INTERVENTIONS:
Device: Footwear — Different types of footwear will be tested to see if these can be used to help slow the progression of osteoarthritis in meniscectomy patients or even stop it from occurring.
  Arms: Meniscus Injured
Procedure: Gait analysis — Gait analysis will be done during several different tasks wear the footwear
  Arms: Footwear

SUMMARY:
Injuries to the meniscus are common in sport. A meniscectomy is often performed to manage symptoms associated with the meniscal injury. Following a meniscectomy individuals are highly likely to develop knee osteoarthritis (OA). Footwear interventions have demonstrated biomechanical changes during walking and running, in healthy and individuals with osteoarthritis. With the increased risk of developing OA associated with meniscectomy patients, understanding biomechanical changes with footwear when compared to healthy individuals, may provide a conservative approach to delaying or minimising the development of (OA). There is no current literature assessing the effect footwear has post meniscectomy, so this is a very novel approach and can yield important results for the management of future risks. Current evidence supports the use of footwear interventions aiming to minimise OA progression in older adults during walking. Yet, meniscectomy patients who have sustained an injury during sport are likely to continue to participate in sport following treatment in their usual footwear. Further evidence is required to better understand the effect of footwear interventions during dynamic movements often performed in sport. Previous studies have assessed customised footwear interventions, however these interventions are not representative of commercially available interventions that could be widely used by the general population. Therefore assessing commercially available footwear will give a more realistic approach to conservative treatment for meniscectomy patients. This project aims to examine biomechanical differences between commercially available footwear conditions in healthy individuals and individuals who have had a meniscal injury. Three-dimensional kinetic and kinematic measures will be assessed during five tasks (walking, running, 90 degrees side cut, single leg landing, and small knee bend squat), for different footwear conditions.

DETAILED DESCRIPTION:
Injuries to the meniscus are common in sport, often as a result of a traumatic event. Mitchell et al. (2016) reported 5.1 meniscal injuries per 100 000 athletic exposures, with a greater proportion reported during competition (11.9 injuries per 100 000 athletic exposures), compared to practice (2.7 injuries per 100 000 athletic exposures). Rotation around a planted/ inverted foot has been cited as a common mechanism for meniscal injuries, followed by landing and jumping movements. The meniscus aids in stabilising the knee, acting as a shock absorber and transmitting load. Damage to the meniscus is suggest to lead to altered knee mechanics leading to the initiation or acceleration of osteoarthritis (OA) development. Prior meniscal tears are commonly reported in OA patients, in addition, reports suggest 4 to 14 times increased risk of developing OA following a meniscal injury.

Altered knee mechanics have been reported following a meniscal injury, which have been associated with increased likelihood of developing OA. These changes include reduced contact area within the joint and increased contact pressure, resulting in reduced ability to transmit load. Indirect measures of knee loading, such as external knee adductor moments (EKAM) and knee adduction angular impulses (KAAI), have been associated with increased risk of developing OA. Knee joint loading is also determined by the coordination of muscle activity. Greater and longer co-contractions of the medial muscles at the knee have demonstrated faster development of OA in individuals diagnosed with medial knee OA.

Meniscectomies are widely used to manage the symptoms associated with meniscus injuries. Whilst, non-operative therapies have demonstrated improvements in knee pain three years post intervention. However, following these interventions, alter mechanics of the knee have been observed. For instance, following a medial meniscectomy, increases in contact area and pressure at the knee have been observed and suggested to increase the likelihood of developing OA. Increases in EKAM in meniscectomy patients have been associated with changes in tibia alignment and GRF lever arm. Non-invasive interventions such as footwear, could alter biomechanics to lower EKAM and reduce the progression of OA. Following a meniscectomy procedure, most patients tend to go back to wearing their old trainers. Due to the changes in the biomechanics of the knee, it can be assumed that they support and cushioning they need would change too.

Typical sports movements such as landing and cutting require dynamic control of the knee which is very under-researched. Muscle strength recovery is also considered to be important for young individuals after an arthroscopic surgery in order to regain capacity to participate in sports or other activities as both pre- and post-operative knee extensor strength have been reported to predict better functional outcome of knee surgery. The co-contraction between the quadriceps and hamstrings are also important in this as muscle weakness creates a less stable base. Muscle strength is also essential to control movements such as stair descent which is essential for everyday living. This is closely linked with balance and the risk of falling. Having extra support or cushioning in footwear can help aid this control needed for static and dynamic exercises especially post-surgical intervention.

Different footwear interventions have been used in OA patients to reduce knee loading and pain. Lateral wedges have demonstrated reduced medial knee loading in both affected and contralateral limbs. In addition, mobility shoes and lateral wedges which provide additional medial support have been shown to reduce pain in OA patients. However, it is unclear whether footwear interventions are able to alleviate the risk factors associated with the progression of OA following a meniscal injury. For effective self-management, post operation the appropriate footwear is recommended, however there is little evidence to inform what the appropriate footwear is for patient after surgery or with knee OA.

Current evidence on footwear interventions on minimising OA development relies on assessment of linear movements such as walking and running. Yet, it is likely that athletes who sustain a meniscal injury would return to sport and therefore be required to perform movements that require a greater demand and muscular control then reported during walking. It is unclear whether footwear interventions are able to alleviate the risk factors associated with the progression of OA following a meniscal injury in a younger athletic population. Understanding knee loading during sport-specific movements and between sports footwear can provide a greater insight to the risk of OA development for athletic populations. Therefore understanding the effect of commercially available footwear interventions knee loading during sport-specific movements could provide a greater insight to the use conservative interventions to reducing the risk of OA development for athletic populations.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 40 years
2. Compete and or play sport a minimum two times a week
3. Able to perform sport specific tasks including running, single leg landing and small knee bend squat
4. Meniscectomy group - has had a meniscectomy surgery following a traumatic meniscal injury during a sporting task.

Exclusion Criteria:

1. History of lower extremity surgeries (other than a meniscectomy) e.g. ACL reconstruction
2. Evidence of knee osteoarthritis development either assessed clinically (based on ACR criteria) or radiographically (Kellgren-Lawrence grade >1)
3. Previous history of traumatic (other than the sustained meniscal injury), inflammatory or infectious pathology in the lower extremity
4. Evidence of ligament laxity

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
Biomechanical analysis using 3D motion capture looking at kinematics and kinetics | Change from Baseline until 1 year
  Knee adduction moment curve (different peaks) will be assessed for differences between conditions.
Electromyography analysis of muscle co-contraction | Change from Baseline until 1 year
  The co-activation of quadriceps and hamstrings will be analysed using EMG. EMG will first be normalized using MVC and then the co-contraction will be analysed.
Biomechanical analysis using 3D motion capture looking at kinematics and kinetics | Change from Baseline until 1 year
  Knee adduction angular impulse (the area under the curve) will be assessed for differences between conditions.

SECONDARY OUTCOMES:
Knee injury and osteoarthritis outcome score (KOOS) | Change from Baseline until 1 year
  The KOOS consists of five subscales; Pain, other symptoms, function in daily living (ADL), function in sport and recreation (Sport/Rec) and knee related quality of life (QOL). A five point Likert scale is employed in the questionnaire, with the last week is taken into consideration when answering the questions. A normalised score is calculated for each sub-scale with a score of 100 indicting no symptoms, whilst 0 indicates extreme symptoms.
Patient-perceived global change in pain | Change from Baseline until 1 year
  Patients-perceived global change in pain will be assessed during the tasks. Participants will be asked to complete the five point Likert scale (1 - much worse, 2 - slightly worse, 3 - no change, 4 - slightly better, 5 - much better) following each task (Hinman et al., 2008).
Tampa Scale of Kinesiophobia (TSK) | Change from Baseline until 1 year
  The TSK is a 17-item questionnaire, which asks individuals to rate the extent to which they agree with statements such as 'pain always means that I injured my body' on a 4-point rating scale, with 1 = strongly disagree and 4 = strongly agree (Nicholas et al., 2008). This is to look at whether any changes in the data are because a participant physically cannot move any different or whether they are subconsciously cautious because they have a fear of pain (Miller, Kori and Todd 1991).
Comfort Rating Questionnaire | Change from Baseline until 1 year
  Differences in the overall comfort of the footwear will be assessed using a 10 cm visual analogue scale (Appendix 9). This measure has been reported to be reliable assessment of comfort (Mündermann et al., 2002). Comfort ratings have been show to detect likelihood of compliance and has been related to injury prevalence (Mündermann et al., 2001).

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester Institute of Health and Performance, Manchester, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The research data will only be shared in the research team participating in this study.

REFERENCES:
- [Derived] Starbuck C, Walters V, Herrington L, Barkatali B, Jones R. Knee Offloading by Patients During Walking and Running After Meniscectomy. Orthop J Sports Med. 2024 Mar 21;12(3):23259671231214766. doi: 10.1177/23259671231214766. eCollection 2024 Mar. PMID 38524891